CLINICAL TRIAL: NCT01349400
Title: Watchful Waiting vs. Repair of Oligosymptomatic Incisional Hernias
Brief Title: Watchful Waiting Versus Repair of Oligosymptomatic Incisional Hernias
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Johannes Lauscher, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS6-233
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Incisional Hernia
Keywords: asymptomatic; minimally symptomatic
MeSH Terms: conditions — Incisional Hernia | interventions — Watchful Waiting; Herniorrhaphy

STUDY DESIGN:
Intervention Model Description: Watchful waiting vs. surgical repair
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- watchful waiting (Experimental): After informed consent and randomization into the watchful waiting group patients will receive standardized verbal information and written instructions on symptoms of acute incarceration. In case of acute symptoms they will be told to visit a physician immediately. On follow-up visits at 1 month, 12 months and 24 months the hernia size will be determined by physical examination, and the pain/ discomfort and the functional status will be monitored.
  Control intervention/ reference test:
  Open or laparoscopic hernia repair with mesh (non-absorbable or partly-absorbable alloplastic material) or with direct suture repair. For hernias measuring ≥ 3 cm mesh repair is recommended. A wide overlap of the mesh over the fascia margin on each side has to be provided. Divergent types of repair are permitted but have to be documented.
  Interventions: Other: Watchful waiting
- Hernia repair (Active Comparator): Intervention: Open or laparoscopic hernia repair with mesh (non-absorbable or partly-absorbable alloplastic material) or with direct suture repair. For hernias measuring ≥ 3 cm mesh repair is recommended. A wide overlap of the mesh over the fascia margin on each side has to be provided. Divergent types of repair are permitted but have to be documented.
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Other: Watchful waiting — Watchful waiting means the observation of the hernia. The patient is informed about signs of deterioration or incarceration. The hernia is controlled clinically on defined follow-up visits.
  Arms: watchful waiting
Procedure: Hernia repair — Open or laparoscopic hernia repair with mesh (non-absorbable or partly-absorbable alloplastic material) or with direct suture repair. For hernias measuring ≥ 3 cm mesh repair is recommended. A wide overlap of the mesh over the fascia margin on each side has to be provided.
  These are all standard techniques in incisional hernia repair.
  Arms: Hernia repair

SUMMARY:
Watchful waiting is non-inferior to surgical repair of asymptomatic and oligosymptomatic incisional hernias in terms of pain and discomfort during normal activities.

DETAILED DESCRIPTION:
Incisional hernias are one of the most frequent complications in abdominal surgery. In Germany, 44.000 incisional hernia repairs per year are performed. Incisional hernia repair is not a low risk operation associated with high recurrence rate and high percentage of postoperative pain. Treatment of incisional hernias represents a significant surgical and socioeconomic problem. Until now, surgical treatment is recommended for patients with incisional hernia independent of symptoms due to the risk of an acute incarceration with serious complications. Studies defining the exact indications for incisional hernia repair and describing the natural course of an incisional hernia including the risk of an acute incarceration are not available to date. Randomized controlled trials having been performed in the past few years show that observation is a reasonable option in mildly symptomatic inguinal hernias. In this study, watchful waiting vs. surgical repair of oligosymptomatic incisional hernias are compared in a prospective-randomized setting for the first time.

The primary endpoint is pain during normal activities measured on the Surgical Pain Scales (SPS) after 24 months follow-up. SPS are a numeric analog scale (NAS) from 0 (no pain) to 150 (maximal pain). The primary endpoint will be dichotomized to no/minimal pain (SPS 0-30) and pain interfering with everyday activities (SPS > 30). Watchful waiting is non-inferior to surgical repair in case the upper border of the 95 % confidence interval will not include the value of 2.

Secondary outcomes are pain and discomfort during during sports, at rest, patient satisfaction, quality of life, and the frequency of incarceration. The investigators hypothesize that pain intensity during everyday activities is not different in the compared groups and that incarceration frequency is low. If this was the case, a watchful waiting strategy could be applied in oligosymptomatic incisional hernias and risks and costs for surgery could be saved.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* asymptomatic/ oligosymptomatic incisional hernia

Exclusion Criteria:

* no hernia detectable by physical examination
* acute incarcerated hernia
* emergency hernia repair
* pain or discomfort associated with the hernia during normal activities
* local or systemic infection
* ASA score >3
* inability to complete or comprehend the preoperative questionnaire
* repair with biologic prothesis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2011-11; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Pain/ discomfort during normal activities | 24 months
  Pain/ discomfort during normal activities as a result of the hernia or hernia operation 2 years after enrolment measured by the hernia-specific Surgical Pain Scale (SPS) on a 150 mm-scale ranging from "no pain sensation" to "most intense pain imaginable".

SECONDARY OUTCOMES:
Patient satisfaction with care (5 point Likert scale) | 24 months
  Patient satisfaction with care is measured by standardized questions by 5 point Likert scale
Pain/discomfort at rest /pain during sports /maximal pain | 24 months
  Pain/ discomfort as a result of hernia / hernia operation; SPS
Pain Disability Index | 24 months
  Limitations of normal activities caused by hernia related pain
Quality of Life (SF-36) | 24 months
  Functional status / quality of life
Frequency of acute incarcerations | 24 months
  Number of acute incacerations in relation to length of watchful waiting

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C Lauscher, M. D., Principal Investigator — Charité Campus Benjamin Franklin, Berlin, Germany
Locations (1):
- Charité Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Lauscher JC, Martus P, Stroux A, Neudecker J, Behrens U, Hammerich R, Buhr HJ, Ritz JP. Development of a clinical trial to determine whether watchful waiting is an acceptable alternative to surgical repair for patients with oligosymptomatic incisional hernia: study protocol for a randomized controlled trial. Trials. 2012 Feb 7;13:14. doi: 10.1186/1745-6215-13-14. PMID 22314130